CLINICAL TRIAL: NCT05976594
Title: Long-term Effectiveness of a Recombinant Hepatitis E Vaccine: a Test-negative Design Study
Brief Title: Long-term Effectiveness of a Recombinant Hepatitis E Vaccine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiamen University (Other)
Collaborators: Dongtai Center for Disease Control and Prevention (Unknown); Dongtai Hospital of Traditional Chinese Medicine (Unknown); Dongtai People's Hospital (Unknown)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Other Study IDs: PRO-HE-004-2
Record Dates: First submitted 2023-07-19; First posted 2023-08-04 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis E
Keywords: Hepatitis E; Test-Negative Design; Effectiveness; Vaccine; Rat hepatitis E virus infection
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Clinical residual serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HE group: Subjects who has been diagnosed as HE.
  Interventions: Diagnostic Test: serology and virology detection of hepatitis E virus
- Control group: Subjects who didn't meet the diagnosis criteria of HE.
  Interventions: Diagnostic Test: serology and virology detection of hepatitis E virus

INTERVENTIONS:
Diagnostic Test: serology and virology detection of hepatitis E virus — Serum will be tested for HEV serology and virology, including HEV-IgM, HEV-IgG, HEV-antigen, and HEV-RNA for HEV species A (HEV-A) and HEV species C (HEV-C)，and further HEV genotyping for those positive for HEV-RNA.

SUMMARY:
This test-negative study is designed to evaluate the long-term effectiveness of hepatitis E vaccine (Hecolin®) and to explore the prevalence of rat hepatitis E in Dongtai City.

DETAILED DESCRIPTION:
In this negative test study, residual clinical serum will be collected from 13 hospitals in Dongtai, if it was from patients born between 1941-1991 from 11 towns in Dongtai, who tested positive for ALT levels higher than 2.5 times the upper limit of normal (ULN). Detection of HEV IgM, IgG, antigen, RNA will be performed to diagnose hepatitis E (HE) in each individual. In addition, HE vaccination history will be collect. All the information above will be used to evaluate the long-term effectiveness of HE vaccine. Based on the study design, virological and serological detection (IgM, IgG, antigen, and RNA) of hepatitis E virus species C (HEV-C) will be performed to analyze the prevalence of rat hepatitis E infection in Dongtai.

ELIGIBILITY:
Inclusion Criteria:

1. From 11 townships（Anfeng、Fuan、Tangyang、Hougang、Liangduo、Qingdong、Shiyan、Shenzao、Wulie、Xuhe、Xinjie）
2. ALT ≥ 2.5 ULN
3. Born between 1941 and 1991

Ages: 32 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the designated township who met the criteria of "ALT ≥ 2.5 ULN" and born between 1941 and 1991 will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Estimated)
Dates: Start 2023-08-12 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of hepatitis E infection | Two months after sampling
  In patients with ALT > 2.5 ULN, HEV infection is diagnosed as positive when two of the following indicators are positive: (1) HEV-IgM; (2) Seroconversion or four-fold increase of HEV-IgG；(3) HEV-RNA; (4) HEV-antigen.

SECONDARY OUTCOMES:
Rate of rat hepatitis E infection | Two months after sampling
  In patients with ALT > 2.5 ULN, rat hepatitis E infection is diagnosed as positive when two of the following virologic or serological tests are positive: (1) IgM anti-HEV-C-; (2) IgG anti-HEV-C- seroconversion or four-fold increase；(3) HEV-C-RNA; (4) HEV-C-antigen.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jun, M.D., Study Director — National Institute of Diagnostics and Vaccine Development in infectious disease, Xiamen University
Locations (1):
- Dongtai Center for Disease Control and Prevention, Dongtai, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Data sharing requires investigator consent

REFERENCES:
- [Background] Zhu FC, Zhang J, Zhang XF, Zhou C, Wang ZZ, Huang SJ, Wang H, Yang CL, Jiang HM, Cai JP, Wang YJ, Ai X, Hu YM, Tang Q, Yao X, Yan Q, Xian YL, Wu T, Li YM, Miao J, Ng MH, Shih JW, Xia NS. Efficacy and safety of a recombinant hepatitis E vaccine in healthy adults: a large-scale, randomised, double-blind placebo-controlled, phase 3 trial. Lancet. 2010 Sep 11;376(9744):895-902. doi: 10.1016/S0140-6736(10)61030-6. Epub 2010 Aug 20. PMID 20728932
- [Background] Zhang J, Zhang XF, Huang SJ, Wu T, Hu YM, Wang ZZ, Wang H, Jiang HM, Wang YJ, Yan Q, Guo M, Liu XH, Li JX, Yang CL, Tang Q, Jiang RJ, Pan HR, Li YM, Shih JW, Ng MH, Zhu FC, Xia NS. Long-term efficacy of a hepatitis E vaccine. N Engl J Med. 2015 Mar 5;372(10):914-22. doi: 10.1056/NEJMoa1406011. PMID 25738667